CLINICAL TRIAL: NCT01199302
Title: A Long-term Assessment of Safety and Efficacy of AMG 827 Treatment in Subjects With Crohn's Disease
Brief Title: Long-term Safety Study of Brodalumab in Adults With Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early based on an imbalance in worsening Crohn's disease in active treatment groups.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20100008; 2010-020881-53 (EudraCT Number)
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Results first posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-11

CONDITIONS: Crohn's Disease
Keywords: Amgen; Crohn's; Inflammatory Bowel Disease; IBD; Irritable Bowel Syndrome; IBS; Inflammation; bowel; colon; gastrointestinal
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Irritable Bowel Syndrome; Inflammation | interventions — brodalumab

ARMS (1):
- Brodalumab 350 mg (Experimental): Participants received brodalumab 350 mg intravenously (IV) on day 1, week 4 and every 4 weeks thereafter for up to 132 weeks.
  Interventions: Biological: Brodalumab

INTERVENTIONS:
Biological: Brodalumab — Administered intravenously once every 4 weeks
  Other Names: AMG 827

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of long-term treatment with brodalumab in adults with Crohn's disease.

DETAILED DESCRIPTION:
This study is an open-label extension of study 20090072 (NCT01150890) in adults with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject was randomized into study 20090072 (NCT01150890) and completed the week 12 evaluation.
* Subject completed the week 12 evaluation in study 20090072 no more than 1 year prior to the planned first visit of AMG 827 in 20100008.
* Subject or subject's legally acceptable representative has provided informed consent.
* Subject meets regional recommendations for immunizations, eg, United States Centers for Disease Control and Prevention recommendations for subjects enrolled in the United States.
* For subjects with ≥ 3 months between the week 12 visit of 20090072 and the planned first dose of AMG 827 in 20100008: If testing is clinically indicated in the opinion of the investigator (eg, because of known recent exposure), then subject has negative test for hepatitis B, hepatitis C, and/or human immunodeficiency virus (HIV).
* For female subjects with ≤ 4 weeks between the week 12 visit of 20090072 and the planned first dose of AMG 827 in 20100008: Subject has a negative urine pregnancy test at baseline prior to the first dose of AMG 827 in the open-label extension (except those at least 2 years post menopausal or surgically sterile).
* For female subjects with > 4 weeks between the week 12 visit of 20090072 and the planned first dose of AMG 827 in 20100008: Subject has a negative serum pregnancy test within 28 days before initiating AMG 827 and a negative urine pregnancy test at baseline prior to the first dose of AMG 827 in the open-label extension (except those at least 2 years post menopausal or surgically sterile).
* For subjects with ≥ 3 months between the week 12 visit of 20090072 and the planned first dose of AMG 827 in 20100008, if clinically indicated in the opinion of the investigator (eg, because of known recent exposure) please assess the following:
* If the subject entered 20090072 with a negative purified protein derivative (PPD) test: Subject must have a negative PPD test within 30 days prior to the planned first dose of AMG 827. Tuberculin skin tests should be considered positive when they have greater than or equal to 5 mm of induration at 48-72 hours after test is placed.
* If the subject entered 20090072 with a positive PPD: Subject must have a negative Quantiferon test within 30 days prior to the planned first dose of AMG 827.

Exclusion Criteria:

* Subject had any serious adverse event reported during study 20090072 and considered to be related to investigational product.
* Subject experienced an adverse event or laboratory abnormality in study 20090072 that, in the opinion of the investigator, could cause extension of treatment to be detrimental to the subject, prevent the subject from completing the study, or interfere with the interpretation of the study results.
* Subject has known sensitivity to any of the products to be administered during dosing.

Other medical conditions

* Subject is currently experiencing an infection of Common Terminology Criteria for Adverse Events grade 2 (if requiring oral medication) or higher. Subject is ineligible until the infection resolves.
* Subject has a serious infection, defined as requiring hospitalization or intravenous antibiotics, within 8 weeks before the first dose of AMG 827 in 20100008.
* For subjects with ≥ 3 months between the week 12 visit of 20090072 and the planned first dose of AMG 827 in 20100008: Subject has recurrent or chronic infections, defined as ≥ 3 infections requiring anti-microbials over the past 12 months prior to screening.
* Subject has a significant concurrent medical condition, including
* Type 1 diabetes
* Uncontrolled type 2 diabetes
* Moderate to severe heart failure (New York Heart Association class III or IV)
* Myocardial infarction within the last year
* Current or history of unstable angina pectoris within the last year
* Uncontrolled hypertension as defined by resting blood pressure ≥ 150/90 mmHg prior to first investigational product dose (confirmed by a repeat assessment)
* Severe chronic pulmonary disease (eg, requiring oxygen therapy)
* Major chronic inflammatory disease or connective tissue disease other than Crohn's disease (eg, systemic lupus erythematosus, rheumatoid arthritis, psoriasis)
* Active malignancy, including evidence of cutaneous basal or squamous cell carcinoma or melanoma
* History of cancer (except successfully treated in situ cervical cancer or squamous or basal cell carcinoma of the skin).
* Any condition that, in the opinion of the investigator, might cause this study to be detrimental to the subject
* Laboratory abnormalities
* For subjects with > 4 weeks between the week 12 visit of 20090072 and the planned first dose of AMG 827 in 20100008, subject has laboratory abnormalities at screening, including
* Elevated aspartate aminotransferase or alanine aminotransferase (> 2x upper limit of normal)
* Serum direct bilirubin ≥ 1.5x upper limit of normal
* Hemoglobin < 10 g/dL
* Hemoglobin A1c > 8.0 (for subjects with type 2 diabetes)
* Platelet count < 125,000 /mm^3
* White blood cell count < 3,000 cells/mm^3
* Absolute neutrophil count < 2,000/mm^3
* Creatinine clearance < 50 mL/min (Cockroft-Gault formula, central lab will calculate value and provide to sites)
* Any other laboratory abnormality, which, in the opinion of the investigator, could cause extension of treatment to be detrimental to the subject, prevent the subject from completing the study, or interfere with the interpretation of the study results
* Washouts and non-permitted drugs
* Subject has used Tysabri (natalizumab) subsequent to study 20090072.
* Subject received an anti-tumor necrosis factor agent within 8 weeks prior to the first dose of AMG 827 in 20100008.
* Subject received other commercially available biologic agent (eg, ustekinumab) within 12 weeks prior to the first dose of AMG 827 in 20100008.
* Subject received an investigational agent (other than AMG 827), investigational procedure, or participated in an investigational device study subsequent to study 20090072.
* Subject received live vaccines within 12 weeks prior to the first dose of AMG 827 in 20100008.
* Subject received cyclosporine, mycophenolate mofetil, sirolimus (rapamycin), thalidomide, or tacrolimus within 4 weeks prior to the first dose of AMG 827 in 20100008.
* General or other
* Female subject is not willing to use highly effective contraception during treatment with AMG 827 (except if at least 2 years postmenopausal or surgically sterile).
* Subject is pregnant or breast feeding, or planning to become pregnant while enrolled in the study.
* Subject has any kind of disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or to comply with all required study procedures.
* Subject will not be available for protocol required study visits, to the best of the subject and investigator's knowledge.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-02-02 (Actual); Primary Completion 2011-10-18 (Actual); Study Completion 2011-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (33):
- United States (11):
  - Research Site, Birmingham, Alabama
  - Research Site, Jacksonville, Florida
  - Research Site, Hammond, Louisiana
  - Research Site, Chevy Chase, Maryland
  - Research Site, Rochester, Minnesota
  - Research Site, Mexico, Missouri
  - Research Site, Great Neck, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, San Antonio, Texas
  - Research Site, Ogden, Utah
- Australia (4):
  - Research Site, Kurralta Park, South Australia
  - Research Site, Box Hill, Victoria
  - Research Site, Fitzroy, Victoria
  - Research Site, Fremantle, Western Australia
- Belgium (4):
  - Research Site, Bonheiden
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Roeselare
- Canada (4):
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Hamilton, Ontario
  - Research Site, Montreal, Quebec
- France (5):
  - Research Site, Lille
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
- Research Site, Amsterdam, Netherlands
- Poland (2):
  - Research Site, Bydgoszcz
  - Research Site, Sopot
- Spain (2):
  - Research Site, Barcelona, Catalonia
  - Research Site, Pontevedra, Galicia

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants who had completed the week 12 visit of the parent study 20090072 (NCT01150890).
  The study was conducted at 28 centers in Australia, Belgium, Canada, Spain, France, Netherlands, Poland, and the United States (US).
Pre-assignment Details: In this long-term open-label extension study participants were to receive brodalumab 350 mg every 4 weeks. Results are reported by treatment group assigned in the parent study.
Groups:
- Placebo / Brodalumab 350 mg: Participants who received placebo in the parent study received brodalumab 350 mg intravenously (IV) every 4 weeks (Q4W) for up to 132 weeks.
- Brodalumab 210 mg / 350 mg: Participants who received 210 mg brodalumab Q4W in the parent study received brodalumab 350 mg IV Q4W for up to 132 weeks.
- Brodalumab 350 mg / 350 mg: Participants who received 350 mg brodalumab Q4W in the parent study received brodalumab 350 mg IV Q4W for up to 132 weeks.
- Brodaluamb 700 mg / 350 mg: Participants who received 700 mg brodalumab Q4W in the parent study received brodalumab 350 mg IV Q4W for up to 132 weeks.
Period: Overall Study
Arm/Group | Placebo / Brodalumab 350 mg | Brodalumab 210 mg / 350 mg | Brodalumab 350 mg / 350 mg | Brodaluamb 700 mg / 350 mg
Started | 20 | 16 | 20 | 11
Completed | 0 | 0 | 0 | 0
Not Completed | 20 | 16 | 20 | 11
Not completed — Adverse Event | 1 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 3 | 0
Not completed — Disease Progression | 3 | 4 | 4 | 2
Not completed — Study Termination | 13 | 8 | 11 | 9
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants who were enrolled and treated with at least one dose of brodalumab in the extension study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo / Brodalumab 350 mg | Brodalumab 210 mg / 350 mg | Brodalumab 350 mg / 350 mg | Brodaluamb 700 mg / 350 mg | Total
Number analyzed (Participants) | 20 | 16 | 20 | 11 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (12.0) | 36.3 (10.0) | 35.4 (13.4) | 37.6 (13.2) | 35.9 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 12 | 7 | 38
  Male | 11 | 6 | 8 | 4 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 18 | 12 | 14 | 10 | 54
  Unknown or Not Reported | 2 | 4 | 5 | 1 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 17 | 11 | 14 | 9 | 51
  Other | 1 | 0 | 1 | 1 | 3
  Unknown | 2 | 4 | 5 | 1 | 12
Crohn's Disease Activity Index (CDAI) at Baseline of Parent Study [Mean (Standard Deviation); unit: score on a scale] — The CDAI measures the severity of active disease using 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). The CDAI score is calculated by summing weighted scores for each item. CDAI scores range from 0 to 600, with higher scores indicating greater disease activity. Population: Participants with available data
  score on a scale
    number analyzed (Participants) | 20 | 15 | 20 | 11 | 66
    (all) | 317.24 (65.21) | 321.13 (54.01) | 336.90 (58.92) | 298.37 (43.75) | 320.94 (57.87)
Crohn's Disease Activity Index (CDAI) at Baseline of Extension Study [Mean (Standard Deviation); unit: score on a scale] — The CDAI measures the severity of active disease using 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). The CDAI score is calculated by summing weighted scores for each item. CDAI scores range from 0 to 600, with higher scores indicating greater disease activity. Population: Participants with available data
  score on a scale
    number analyzed (Participants) | 19 | 14 | 19 | 11 | 63
    (all) | 257.70 (126.60) | 251.72 (85.23) | 233.50 (110.74) | 226.76 (65.49) | 243.67 (102.89)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial subject including worsening of a pre-existing medical condition, and not necessarily having a causal relationship with study treatment. A treatment-emergent AE is an event that occurred after the initiation of study drug or was already present prior to the initiation of study drug but worsened in either intensity or frequency after the initiation of study drug.
  The investigator assessed whether each AE was possibly related to the study drug.
  A serious adverse event is defined as an AE that met at least 1 of the following serious criteria:
  * fatal,
  * life threatening,
  * required in-patient hospitalization or prolongation of existing hospitalization,
  * resulted in persistent or significant disability/incapacity,
  * congenital anomaly/birth defect, and/or
  * other significant medical hazard.
Time Frame: From first dose of study drug until the end of study; median (min, max) duration was 70 days (14, 223)
Population: All enrolled participants who received at least one dose of brodalumab in the extension study
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo / Brodalumab 350 mg | Brodalumab 210 mg / 350 mg | Brodalumab 350 mg / 350 mg | Brodaluamb 700 mg / 350 mg
Number analyzed (Participants) | 20 | 16 | 20 | 11
Participants
  All treatment-emergent adverse events (TEAEs) | 14 | 12 | 18 | 8
  Serious adverse events | 4 | 4 | 5 | 2
  Fatal adverse events | 0 | 0 | 0 | 0
  TEAEs leading to discontinuation of study drug | 4 | 1 | 3 | 1
  TEAEs leading to discontinuation from study | 3 | 2 | 3 | 1
  Treatment-related treatment-emergent adverse events | 8 | 9 | 14 | 2
  Treatment-related serious adverse events | 2 | 2 | 1 | 1
  Treatment-related fatal adverse events | 0 | 0 | 0 | 0
  Treatment-related TEAEs leading to discontinuation of study drug | 2 | 1 | 1 | 0
  Treatment related TEAEs leading to discontinuation from study | 1 | 1 | 1 | 0

2. Primary Outcome: Percentage of Participants Who Achieved a CDAI Response
Description: CDAI response is defined as a reduction from baseline in CDAI score of ≥ 100 points.
  The CDAI measures the severity of active disease using 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). The CDAI score is calculated by summing weighted scores for each item. CDAI scores range from 0 to 600, with higher scores indicating greater disease activity.
Time Frame: Baseline of the parent study and weeks 2, 4, 6, 8, 10, 12, 16, and 20
Population: Participants in the full analysis set with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo / Brodalumab 350 mg | Brodalumab 210 mg / 350 mg | Brodalumab 350 mg / 350 mg | Brodaluamb 700 mg / 350 mg
Number analyzed (Participants) | 20 | 16 | 20 | 11
percentage of participants
  Week 2: number analyzed (Participants) | 17 | 14 | 18 | 11
  Week 2 | 23.5 | 21.4 | 50.0 | 54.5
  Week 4: number analyzed (Participants) | 13 | 11 | 19 | 9
  Week 4 | 23.1 | 36.4 | 47.4 | 55.6
  Week 6: number analyzed (Participants) | 13 | 9 | 15 | 7
  Week 6 | 38.5 | 33.3 | 53.3 | 42.9
  Week 8: number analyzed (Participants) | 10 | 7 | 15 | 6
  Week 8 | 40.0 | 42.9 | 40.0 | 83.3
  Week 10: number analyzed (Participants) | 8 | 5 | 11 | 4
  Week 10 | 62.5 | 20.0 | 27.3 | 100.0
  Week 12: number analyzed (Participants) | 6 | 4 | 8 | 5
  Week 12 | 83.3 | 25.0 | 62.5 | 80.0
  Week 16: number analyzed (Participants) | 4 | 0 | 3 | 2
  Week 16 | 100.0 |  | 33.3 | 100.0
  Week 20: number analyzed (Participants) | 4 | 1 | 1 | 2
  Week 20 | 100.0 | 0.0 | 100.0 | 50.0

3. Primary Outcome: Percentage of Participants Who Achieved Clinical Remission
Description: Clinical remission is defined by a CDAI score of ≤ 150 points. The CDAI measures the severity of active disease using 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). The CDAI score is calculated by summing weighted scores for each item. CDAI scores range from 0 to 600, with higher scores indicating greater disease activity.
Time Frame: Weeks 2, 4, 6, 8, 10, 12, 16, and 20
Population: Participants in the full analysis set with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo / Brodalumab 350 mg | Brodalumab 210 mg / 350 mg | Brodalumab 350 mg / 350 mg | Brodaluamb 700 mg / 350 mg
Number analyzed (Participants) | 20 | 16 | 20 | 11
percentage of participants
  Week 2: number analyzed (Participants) | 17 | 14 | 18 | 11
  Week 2 | 5.9 | 7.1 | 27.8 | 27.3
  Week 4: number analyzed (Participants) | 13 | 11 | 19 | 9
  Week 4 | 15.4 | 9.1 | 26.3 | 22.2
  Week 6: number analyzed (Participants) | 13 | 9 | 15 | 7
  Week 6 | 23.1 | 0.0 | 33.3 | 28.6
  Week 8: number analyzed (Participants) | 10 | 7 | 15 | 6
  Week 8 | 40.0 | 0.0 | 13.3 | 50.0
  Week 10: number analyzed (Participants) | 8 | 5 | 11 | 4
  Week 10 | 37.5 | 0.0 | 18.2 | 75.0
  Week 12: number analyzed (Participants) | 6 | 4 | 8 | 5
  Week 12 | 50.0 | 0.0 | 50.0 | 60.0
  Week 16: number analyzed (Participants) | 4 | 0 | 3 | 2
  Week 16 | 75.0 |  | 33.3 | 0.0
  Week 20: number analyzed (Participants) | 4 | 1 | 1 | 2
  Week 20 | 100.0 | 0.0 | 100.0 | 0.0

4. Secondary Outcome: CDAI Score Over Time
Description: The CDAI measures the severity of active disease using 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). The CDAI score is calculated by summing weighted scores for each item. CDAI scores range from 0 to 600, with higher scores indicating greater disease activity.
Time Frame: Weeks 2, 4, 6, 8, 10, 12, 16, and 20
Population: Participants in the full analysis set with available data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo / Brodalumab 350 mg | Brodalumab 210 mg / 350 mg | Brodalumab 350 mg / 350 mg | Brodaluamb 700 mg / 350 mg
Number analyzed (Participants) | 20 | 16 | 20 | 11
score on a scale
  Week 2: number analyzed (Participants) | 17 | 14 | 18 | 11
  Week 2 | 291.71 (159.01) | 285.41 (86.69) | 235.12 (100.66) | 197.71 (81.22)
  Week 4: number analyzed (Participants) | 13 | 11 | 19 | 9
  Week 4 | 274.21 (154.79) | 244.11 (62.60) | 256.22 (125.24) | 192.04 (54.62)
  Week 6: number analyzed (Participants) | 13 | 9 | 15 | 7
  Week 6 | 257.09 (154.96) | 274.48 (93.41) | 241.13 (134.06) | 219.91 (121.19)
  Week 8: number analyzed (Participants) | 10 | 7 | 15 | 6
  Week 8 | 250.95 (167.25) | 248.03 (70.86) | 267.51 (173.20) | 159.39 (66.53)
  Week 10: number analyzed (Participants) | 8 | 5 | 11 | 4
  Week 10 | 196.56 (157.07) | 274.81 (90.70) | 276.37 (138.48) | 127.57 (46.38)
  Week 12: number analyzed (Participants) | 6 | 4 | 8 | 5
  Week 12 | 120.47 (93.27) | 317.49 (27.14) | 224.79 (131.61) | 159.91 (61.03)
  Week 16: number analyzed (Participants) | 4 | 0 | 3 | 2
  Week 16 | 103.61 (48.60) |  | 220.67 (178.45) | 186.11 (10.05)
  Week 20: number analyzed (Participants) | 4 | 1 | 1 | 2
  Week 20 | 101.60 (62.32) | 212.42 | 145.33 | 223.11 (13.52)

5. Secondary Outcome: Change From Baseline in CDAI Score Over Time
Description: as for outcome 4
Time Frame: Baseline of the parent study and Weeks 2, 4, 6, 8, 10, 12, 16, and 20
Population: Participants in the full analysis set with available data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo / Brodalumab 350 mg | Brodalumab 210 mg / 350 mg | Brodalumab 350 mg / 350 mg | Brodaluamb 700 mg / 350 mg
Number analyzed (Participants) | 20 | 16 | 20 | 11
score on a scale
  Week 2: number analyzed (Participants) | 17 | 14 | 18 | 11
  Week 2 | -25.8 (128.0) | -35.0 (90.8) | -97.0 (106.9) | -100.7 (83.7)
  Week 4: number analyzed (Participants) | 13 | 11 | 19 | 9
  Week 4 | -49.7 (112.5) | -79.2 (67.6) | -78.2 (107.3) | -101.1 (62.0)
  Week 6: number analyzed (Participants) | 13 | 9 | 15 | 7
  Week 6 | -55.4 (101.4) | -51.5 (106.7) | -84.3 (128.3) | -67.8 (127.6)
  Week 8: number analyzed (Participants) | 10 | 7 | 15 | 6
  Week 8 | -48.7 (143.2) | -84.6 (79.8) | -55.4 (157.2) | -150.4 (35.6)
  Week 10: number analyzed (Participants) | 8 | 5 | 11 | 4
  Week 10 | -116.1 (103.5) | -45.3 (81.5) | -56.1 (146.5) | -182.6 (32.7)
  Week 12: number analyzed (Participants) | 6 | 4 | 8 | 5
  Week 12 | -174.5 (76.0) | -20.7 (69.1) | -80.8 (120.4) | -160.2 (50.3)
  Week 16: number analyzed (Participants) | 4 | 0 | 3 | 2
  Week 16 | -162.1 (51.3) |  | -55.9 (155.5) | -128.8 (33.6)
  Week 20: number analyzed (Participants) | 4 | 1 | 1 | 2
  Week 20 | -164.1 (53.8) | -61.3 | -109.7 | -91.8 (57.2)

6. Secondary Outcome: Number of Participants Who Developed Anti-brodalumab Binding Antibodies
Description: Binding antibodies to brodalumab were detected using an anti-brodalumab immunoassay.
Time Frame: Blood samples were collected at study entry, week 4, 24 and at last visit (maximum time on study was 32 weeks).
Population: Enrolled participants who received at least one dose of brodalumab in the extension study and with available antibody results
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo / Brodalumab 350 mg | Brodalumab 210 mg / 350 mg | Brodalumab 350 mg / 350 mg | Brodaluamb 700 mg / 350 mg
Number analyzed (Participants) | 20 | 16 | 20 | 11
Participants | 0 | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP) Levels Over Time
Time Frame: Baseline of the parent study and Weeks 2, 4, 6, 8, 10, 12, 16, and 20
Population: Participants in the full analysis set with available data at each time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo / Brodalumab 350 mg | Brodalumab 210 mg / 350 mg | Brodalumab 350 mg / 350 mg | Brodaluamb 700 mg / 350 mg
Number analyzed (Participants) | 20 | 16 | 20 | 11
mg/dL
  Week 2: number analyzed (Participants) | 19 | 15 | 18 | 11
  Week 2 | 13.0 (33.9) | 10.7 (53.8) | -3.5 (22.9) | 3.2 (19.8)
  Week 4: number analyzed (Participants) | 15 | 12 | 19 | 10
  Week 4 | -0.8 (9.9) | -0.8 (17.9) | -8.1 (25.9) | 9.9 (52.4)
  Week 6: number analyzed (Participants) | 15 | 9 | 15 | 7
  Week 6 | 5.2 (14.1) | 5.9 (26.2) | -5.1 (30.0) | 17.5 (25.9)
  Week 8: number analyzed (Participants) | 12 | 9 | 15 | 8
  Week 8 | 15.5 (49.2) | -2.4 (15.0) | 3.7 (19.9) | 7.2 (49.5)
  Week 10: number analyzed (Participants) | 9 | 5 | 11 | 4
  Week 10 | 11.5 (31.9) | 4.3 (28.8) | 0.9 (34.1) | -1.2 (2.3)
  Week 12: number analyzed (Participants) | 7 | 5 | 10 | 6
  Week 12 | 2.9 (9.7) | 1.2 (19.1) | 15.4 (34.9) | -11.5 (17.9)
  Week 16: number analyzed (Participants) | 4 | 1 | 3 | 3
  Week 16 | 1.0 (18.1) | 0.2 | -9.5 (11.5) | -15.0 (23.5)
  Week 20: number analyzed (Participants) | 5 | 1 | 1 | 4
  Week 20 | -3.0 (3.4) | -3.2 | -1.1 | -10.9 (21.1)

ADVERSE EVENTS:
Time Frame: From first dose of study drug until the end of study; median (min, max) duration was 70 days (14, 223)
Groups:
- Brodalumab 350 mg Q4W: Participants received brodalumab 350 mg IV Q4W for up to 132 weeks.
Arm/Group | Brodalumab 350 mg Q4W
Serious Adverse Events (participants affected / at risk) | 15/67
Other Adverse Events (participants affected / at risk) | 36/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brodalumab 350 mg Q4W (N=67)
Abdominal pain (Gastrointestinal disorders) | 2
Anal stenosis (Gastrointestinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 7
Intestinal dilatation (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 3
Gastroenteritis (Infections and infestations) | 1
Peritoneal abscess (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brodalumab 350 mg Q4W (N=67)
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal tenderness (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Crohn's disease (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Chills (General disorders) | 3
Fatigue (General disorders) | 5
Pyrexia (General disorders) | 9
Oral candidiasis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Headache (Nervous system disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.